CLINICAL TRIAL: NCT01053416
Title: 10-year Follow up of Patients With Pigment Dispersion Syndrome: Risk Factors for Conversion to Pigmentary Glaucoma and Potential Protective Effect of a Yag-laser Iridotomy in High Risk Eye
Brief Title: Pigment Dispersion Syndrome: Natural History and Possible Protective Effect of a YAG Laser Iridotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: STEFANO A. GANDOLFI, PROFESSOR OF OPHTHALMOLOGY AND CHAIRMAN, UNIVERSITY OF PARMA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PARMAPIGMO
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2003-01

CONDITIONS: Pigment Dispersion Syndrome
Keywords: glaucoma; pigmentary glaucoma; laser iridotomy
MeSH Terms: conditions — Glaucoma-Related Pigment Dispersion Syndrome; Glaucoma; Glaucoma, Open-Angle | interventions — Iridectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- observation (No Intervention)
- Yag laser iridotomy (Experimental): the enrolled eyes will undergo an iridotomy performed by using a Yag-laser
  Interventions: Procedure: Yag laser iridotomy

INTERVENTIONS:
Procedure: Yag laser iridotomy — the procedure will be performed by using a Yag laser. Single spot, 1 mJ power, beam aimed to an existing iris crypt
  Other Names: iridectomy
  Arms: Yag laser iridotomy

SUMMARY:
STUDY AIMS

1. To determine the 10-year conversion rate from pigment dispersion syndrome (PDS) to pigmentary glaucoma (PG)
2. To evaluate the possible protective effect of a Yag-laser iridotomy

DETAILED DESCRIPTION:
1154 workers in the Parma area will be screened for eligibility to long-term use of video-monitors. Those referred to the Glaucoma Clinic for suspected PDS will be enrolled in the study.

In a prospective study on the natural history of PDS and PG, Richter et al. (Arch Ophtal 104:211-5, 1986) found an association between "active pigment dispersion" and elevated IOP. Therefore, in order to evaluate the "stability" of the pigment, a phenylephrine test will be performed following the method reported by Epstein et al (1978) AJO 85:43-50. The test will be performed by one investigator (SAG)and was considered positive if > "grade 1+" (i.e. at least 10 particles in a single light beam). Eyes showing a positive test will be considered as "high-risk" for conversion to PG.

Yag laser iridotomy will be performed in patients showing both eyes at high risk. One eye only (randomly chosen) will be treated. the fellow eye will be left untreated and considered as internal control.

Low risk eyes will be followed without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Krukenberg spindle
* Slit-like mid peripheral iris defect
* Pigment in > 270° of AC angle

Exclusion Criteria:

* IOP > 18 mmHg
* PEX (full mydriasis)
* w/w field defect (Octopus G1 program)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 1993-01; Primary Completion 2003-04 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
> 5 mmHg IOP increase vs baseline (average 2 highest readings, 8 am - 6 pm phasing, 6 readings) | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sezione Di Oftalmologia, Universita' Di Parma, Parma, Italy

REFERENCES:
- [Derived] Gandolfi SA, Ungaro N, Tardini MG, Ghirardini S, Carta A, Mora P. A 10-year follow-up to determine the effect of YAG laser iridotomy on the natural history of pigment dispersion syndrome: a randomized clinical trial. JAMA Ophthalmol. 2014 Dec;132(12):1433-8. doi: 10.1001/jamaophthalmol.2014.3291. PMID 25188224